CLINICAL TRIAL: NCT02214095
Title: Glucosamine Sulphate as an Adjunctive Therapy to Closed Mechanical Debridement Reduced Gingival Cervicular Fluid IL-1β in Patients With Chronic Periodontitis
Brief Title: Glucosamine Periodontal Adjunctive Therapy
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: had been finished
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mai Shafik Attia, lecturer of oral medicine and periodontology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: randomized clinical trial
Record Dates: First submitted 2014-07-08; First posted 2014-08-12 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Periodontitis
Keywords: Cytokines; interleukin-1β; chronic periodontitis; host modulation; glucosamine sulphate.
MeSH Terms: conditions — Chronic Periodontitis | interventions — Glucosamine; Lactose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- glucosamine sulphate capsules (Active Comparator): 500 mg Glucosamine Compound, three times daily for 3 months following initial cause related therapy.
  Interventions: Drug: glucosamine sulphate
- lactose capsules (Placebo Comparator): lactose capsules three times daily for 3 months
  Interventions: Drug: lactose capsules

INTERVENTIONS:
Drug: glucosamine sulphate — group I (G1) patients received 500 mg glucosamine sulphate capsules (Glucosamine Compound) , three times daily for 3 months following initial cause related therapy. Group II patients were given placebo capsules( Lactose) for the same period following initial cause related therapy
  Other Names: antiarthritis drugs; antiinflammatory drugs
  Arms: glucosamine sulphate capsules
Drug: lactose capsules
  Arms: lactose capsules

SUMMARY:
This study is the first evidence based work evaluated the systemic use of glucosamine as an adjunctive therapy to closed mechanical debridement in chronic periodontitis. The use of glucosamine sulphate was correlated with clinical outcomes and IL1-β level in the GCF of patients with moderate to advanced chronic periodontitis

DETAILED DESCRIPTION:
Targeting the inflammatory response may be a rational approach to the medical treatment of chronic periodontitis. Glucosamine sulphate (GS) was proven to have anti-inflammatory actions with minimal side effect profile. Objectives; The main objectives of this study were to evaluate clinically the efficacy of GS; as a novel adjunctive host modulating agent in periodontal therapy and to investigate its effect on gingival crevicular fluid (GCF) level of IL-1β. Methods; Forty patients with moderate to severe chronic periodontitis (CP) were included in this study. They were randomly divided into two groups. Group I (G1) patients (n=20) received 500 mg GS capsules three times daily for 3 months following full mouth scaling and root planing (SRP), while group II (G2) patients (n=20) received a placebo for the same period following full mouth SRP. Clinical periodontal parameters and GCF IL-1β levels were analyzed at baseline and 3 months following therapy.

ELIGIBILITY:
Inclusion Criteria:

1. good compliance with the plaque control instructions following initial therapy
2. each subject contributed a single premolar or molar tooth with interproximal probing depth ≥ 5 mm and clinical attachment loss ≥ 4 mm
3. teeth involved were all vital with score 0-1 mobility
4. availability for the follow-up and maintenance program;

Exclusion Criteria:

1. no systemic diseases which could influence the outcome of therapy as evidenced by Burket's Oral Medicine health history questionnaire
2. absence of periodontal treatment for the previous year
3. absence of systemic medication or antibiotic treatment for the previous six months
4. absence of a smoking habit.
5. post menopausal, pregnant or breast feeding women were excluded from participating in the study. Patients with contraindications to glucosamine sulphate therapy e.g., hypersensitivity to any of the product's components or with inadequate compliance with the oral hygiene maintenance schedule were also excluded from the study.

Ages: 35 Years to 48 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
gingival crevicular fluid IL-1β level | 0-3 months
  baseline and after three months of Glucosamine Sulphate administration

SECONDARY OUTCOMES:
probing depth | 0-3 months
  the distance from the gingival margin to the base of the pocket was measured at baseline and 3 months after drug administration
clinical attachment level | 0-3 months
  distance from cemento-enamel junction and base of the pocket was measured at baseline and 3 months after drug administration
gingival index | 0-3 months
  gingival inflammation was measured by gingival index at baseline and 3 months after drug administration.
plaque index | 0-3 months
  plaque deposits was measured by plaque index at baseline and 3 months after drug therapy

CONTACTS AND LOCATIONS:
Overall Officials: Ahmaed Y Gamal, Principal Investigator — Ainshams University; Hala A Elela, professer, Principal Investigator — Ainshams University; Mai S Attia, Lecturer, Principal Investigator — Al-Azhar University
Locations (1):
- Ainshams University, Cairo, Egypt